CLINICAL TRIAL: NCT05990088
Title: Comparison of Electromyographic Muscle Activity and Occlusal Accuracy Between Conventional and CAD/CAM Complete Dentures Designed Based on Neutral Zone Concept (Randomized Controlled Clinical Trial)
Brief Title: Comparison Between Conventional and CAD/CAM Complete Dentures Designed Based on Neutral Zone Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia M. Refai, Lecturer of Oral and Maxillofacial Prosthodontics, Faculty of Dentistry, Ain Shams Univeristy, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-ReclR012317
Record Dates: First submitted 2023-07-22; First posted 2023-08-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Missing Teeth; Dentures
Keywords: CAD-CAM; Denture, Complete; Electromyography
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat Cured Conventional Complete Removable Dentures based on neutral zone concept (Experimental): The patient will be provided by a complete removable denture designed based on the neutral zone concept to restore his missing teeth which will be manufactured by heat curing of Polymethyl methacrylate.
  Interventions: Device: Heat Cured Conventional Polymethylmethacrylate Complete Removable Dentures based on neutral zone concept
- CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept. (Active Comparator): The patient will be provided with a complete removable denture designed according to the neutral-concept to restore his missing teeth, which will be manufactured by CAD/CAM milling of monolithic methacrylate blanks.
  Interventions: Device: CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept.

INTERVENTIONS:
Device: Heat Cured Conventional Polymethylmethacrylate Complete Removable Dentures based on neutral zone concept — The patients will receive complete removable dentures designed based on neutral zone concept and manufactured by heat cured conventional technique of polymethylmethacrylate
  Arms: Heat Cured Conventional Complete Removable Dentures based on neutral zone concept
Device: CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept. — The patients will receive complete removable dentures designed based on the neutral-zone concept and digitally manufactured using a milling machineز
  Arms: CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept.

SUMMARY:
A within-subject cross-over study is done on eight completely edentulous patients to compare two different complete removable dentures. Group I: Heat cured Conventional complete dentures designed based on the neutral zone concept; Group II: CAD-CAM neutral zone complete dentures designed based on the neutral zone concept. Occlusal analysis is done by the T-Scan device, and evaluation of muscle activity is conducted by electromyography at insertion time, two weeks after insertion time, and one month after insertion time.

DETAILED DESCRIPTION:
This study is designed as a randomized clinical trial applying a within-subject comparison of two different complete denture types as follows; group I: Heat cured Conventional complete dentures designed based on the neutral zone concept, group II: CAD-CAM neutral zone complete dentures designed based on the neutral zone concept. The study will be carried out on eight completely edentulous patients, each patient will receive two sets of complete dentures in a random sequence. For each denture set, at the denture insertion visit occlusal analysis and equilibration will be performed with the aid of the T-Scan device, also EMG evaluation of muscle activity will be conducted. Two weeks after, the patients will be recalled to reanalyze the occlusion after the denture settles using the T-scan computerized system. One month after the last recall visit, the EMG evaluation of muscle activity will be conducted again. The EMG and T-scan recording data will be collected and analyzed to compare the two denture types

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been completely edentulous in both jaws (maxilla and mandible) for a long period.
2. Patients with a resorbed mandibular ridge.
3. Patients with a Class I maxillo-mandibular relationship
4. Patients with adequate inter-arch space.
5. Patients with good neuromuscular control.
6. Patients without any tempo-mandibular disorder.

Exclusion Criteria:

1. Patients with any oral diseases that may affect complete denture construction
2. Patients with bad oral hygiene.
3. Patients with neuromuscular disorders.
4. Patients with a history of parafunctional habits.
5. Hysterical patients.
6. Patients will undergo or have previously received chemotherapy or radiotherapy.
7. Drug-addicted patients.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the electromyography muscle activity (EMG) of the masseter and temporalis muscles. | one month
  The electromyography activity of the Masseter and Temporalis muscles will be evaluated during clenching, chewing of soft food, and chewing of hard food, at the time of denture insertion (baseline) and one month after baseline.The measuring unit is mv.

SECONDARY OUTCOMES:
Evaluation of occlusal force equilibration using t-scan device | two weeks
  The percentage of occlusal force distribution will be evaluated for both dentures using the T-Scan computerized occlusal analysis system, at the time of denture insertion (baseline) and following baseline by two weeks after.

CONTACTS AND LOCATIONS:
Overall Officials: Omnia MS Refai, PHD, Principal Investigator — Faculty of Dentistry Ain Shams University; Omar A El-Sadat, PHD, Principal Investigator — Faculty of Dentistry Ain Shams University; Sara IS Mohamed, PHD, Principal Investigator — Faculty of Dentistry , Ain Shams Univeristy
Locations (1):
- Faculty of Dentistry, Ain shams University, Cairo, Egypt

REFERENCES:
- [Background] Ohkubo C, Shimpo H, Tokue A, Park EJ, Kim TH. Complete denture fabrication using piezography and CAD-CAM: A clinical report. J Prosthet Dent. 2018 Mar;119(3):334-338. doi: 10.1016/j.prosdent.2017.04.013. Epub 2017 Jul 15. PMID 28720338
- [Result] Cagna DR, Massad JJ, Schiesser FJ. The neutral zone revisited: from historical concepts to modern application. J Prosthet Dent. 2009 Jun;101(6):405-12. doi: 10.1016/S0022-3913(09)60087-1. PMID 19463668